CLINICAL TRIAL: NCT04081103
Title: A Phase 2, Randomized, Prospective, Double-masked, Vehicle-controlled Study to Assess the Efficacy and Safety of Nexagon® (NEXAGON) in Subjects With Corneal Persistent Epithelial Defects
Brief Title: NEXAGON for the Treatment of Corneal Persistent Epithelial Defects Following Severe Ocular Injuries
Acronym: EXPEDE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped early (n=35) enabling the data to guide design of the subsequent clinical study.
Sponsor: Glaukos Corporation (Industry)
Collaborators: Amber Ophthalmics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEX-PED-005
Record Dates: First submitted 2019-08-29; First posted 2019-09-09 (Actual); Results first posted 2024-10-23 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Corneal Persistent Epithelial Defect

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Nexagon® (lufepirsen) High Dose Concentration (Experimental)
  Interventions: Drug: Nexagon® (lufepirsen) High Dose Concentration; Drug: Open-label Nexagon® (lufepirsen)
- Nexagon® (lufepirsen) Low Dose Concentration (Experimental)
  Interventions: Drug: Nexagon® (lufepirsen) Low Dose Concentration; Drug: Open-label Nexagon® (lufepirsen)
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle; Drug: Open-label Nexagon® (lufepirsen)

INTERVENTIONS:
Drug: Nexagon® (lufepirsen) High Dose Concentration — Nexagon® (lufepirsen) is administered topically in the affected eye three (3) times over 28 days.
  Arms: Nexagon® (lufepirsen) High Dose Concentration
Drug: Nexagon® (lufepirsen) Low Dose Concentration — Nexagon® (lufepirsen) is administered topically in the affected eye three (3) times over 28 days.
  Arms: Nexagon® (lufepirsen) Low Dose Concentration
Drug: Vehicle — Vehicle is administered topically in the affected eye three (3) times over 28 days.
  Other Names: Placebo
  Arms: Vehicle
Drug: Open-label Nexagon® (lufepirsen) — Open-label Nexagon® (lufepirsen) for participants who do not heal (re-epithelialize) at the end of the 28-day treatment phase.

SUMMARY:
This study will enroll participants with a non-infected, corneal persistent epithelial defect (PED) resulting from an ocular chemical and/or thermal ocular injury which is non-responsive or refractory to current standard of care for at least 14 days. It will assess the efficacy and safety of Nexagon® (lufepirsen) plus standard of care versus NEXAGON-vehicle (placebo) plus standard of care. The recovery of the corneal epithelium will be the primary outcome measure, defined as a cornea that re-epithelializes by Day 28 of treatment and remains re-epithelialized for at least a further 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female of any age.
2. The presence of a non-infected, corneal persistent epithelial defect (PED) which has resulted from a severe chemical and/or thermal (burn) injury to one or both eyes.
3. The PED is non-responsive to current standard of care for at least 14 days from injury.
4. The PED measures at least 2 mm along the largest diameter at Day 1 of the Treatment Period.
5. Providing written informed consent and ability to comply with the visit and dosing schedule.

Exclusion Criteria:

1. Have active ocular infection.
2. Subjects with corneal perforation or impending corneal perforation.
3. Subjects with any other past or present ophthalmic disease or medical condition that, in the Investigator's opinion, may affect the safety of the subject or the outcome of the study.
4. Subjects with severe lid abnormalities or ocular conditions that contribute to the persistence of the epithelial defect.
5. Female subjects of childbearing potential who are pregnant, nursing, planning a pregnancy or not using an adequate and medically acceptable form of birth control.
6. Subjects who have participated in an interventional clinical trial within 30 days prior to Day 1.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Feldman, Study Director — Amber Ophthalmics
Locations (1):
- Jules Stein Eye Institute, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | Nexagon® (Lufepirsen) High Dose Concentration | Nexagon® (Lufepirsen) Low Dose Concentration | Vehicle
Started | 12; 12 Eyes | 12; 12 Eyes | 11; 11 Eyes
Completed | 11; 11 Eyes | 11; 11 Eyes | 9; 9 Eyes
Not Completed | 1; 1 Eyes | 1; 1 Eyes | 2; 2 Eyes
Not completed — Adverse Event | 1 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nexagon® (Lufepirsen) High Dose Concentration | Nexagon® (Lufepirsen) Low Dose Concentration | Vehicle | Total
Number analyzed (Participants) | 12 | 12 | 11 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.9 (20.42) | 30.3 (16.38) | 30.9 (19.03) | 29.0 (18.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 3 | 7
  Male | 9 | 11 | 8 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 11 | 12 | 11 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 11 | 11 | 11 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 1 | 0 | 0 | 1
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 0 | 2
  India | 11 | 11 | 11 | 33
Subjects with of Persistent Epithelial Defect [Count of Participants; unit: Participants] | 12 | 12 | 11 | 35

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects Achieving Corneal Epithelial Recovery, as Assessed by Slit Lamp Examination.
Description: Corneal epithelial recovery, defined as corneal reepithelialization and maintenance of a durable epithelium for at least 28 days, will be assessed by slit lamp examination.
Time Frame: Up to 56 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Nexagon® (Lufepirsen) High Dose Concentration | Nexagon® (Lufepirsen) Low Dose Concentration | Vehicle
Number analyzed (Participants) | 12 | 12 | 11
Participants | 8 | 8 | 3

2. Primary Outcome: Incidence of Treatment Emergent Adverse Events as Assessed by CTCAE v 5.0
Description: Incidence of Treatment Emergent Adverse Events as assessed by CTCAE v 5.0.
Time Frame: Up to 30 days after last application of intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Nexagon® (Lufepirsen) High Dose Concentration | Nexagon® (Lufepirsen) Low Dose Concentration | Vehicle
Number analyzed (Participants) | 12 | 12 | 11
Participants | 7 | 8 | 7

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Nexagon® (Lufepirsen) High Dose Concentration | Nexagon® (Lufepirsen) Low Dose Concentration | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/12 | 0/11
Other Adverse Events (participants affected / at risk) | 7/12 | 8/12 | 7/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nexagon® (Lufepirsen) High Dose Concentration (N=12) | Nexagon® (Lufepirsen) Low Dose Concentration (N=12) | Vehicle (N=11)
Cicatricial ectropion with lateral lagophthalmos and exposed lacrimal gland (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — Study Eye
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nexagon® (Lufepirsen) High Dose Concentration (N=12) | Nexagon® (Lufepirsen) Low Dose Concentration (N=12) | Vehicle (N=11)
Symblepharon (Eye disorders) | 1 | 2 | 3 — Study Eye
Corneal epithelium defect (Eye disorders) | 1 | 0 | 3 — Study Eye
Eye pain (Eye disorders) | 1 | 1 | 0 — Study Eye
Blepharitis (Eye disorders) | 1 | 0 | 0 — Study Eye
Cataract (Eye disorders) | 1 | 0 | 0 — Study Eye
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 1 — Study Eye
Corneal neovascularisation (Eye disorders) | 0 | 1 | 0 — Study Eye
Corneal thinning (Eye disorders) | 1 | 0 | 0 — Study Eye
Dry eye (Eye disorders) | 0 | 1 | 0 — Study Eye
Ectropion (Eye disorders) | 0 | 1 | 0 — Study Eye
Eye irritation (Eye disorders) | 0 | 1 | 0 — Study Eye
Eye pruritus (Eye disorders) | 0 | 1 | 0 — Study Eye
Lacrimation increased (Eye disorders) | 0 | 1 | 0 — Study Eye
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 — Study Eye
Visual impairment (Eye disorders) | 0 | 1 | 0 — Study Eye
Hyperplasia (General disorders) | 0 | 0 | 1 — Study Eye
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 — Study Eye
Hypopyon (Infections and infestations) | 1 | 1 | 1 — Study Eye
Periorbital cellulitis (Infections and infestations) | 0 | 1 | 0 — Study Eye
Eyelid scar (Injury, poisoning and procedural complications) | 1 | 0 | 0 — Study Eye
Cataract (Eye disorders) | 1 | 0 | 0 — Fellow Eye
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 — Fellow Eye
COVID-19 (Infections and infestations) | 0 | 1 | 0 — Non-Ocular
Blood bilirubin increased (Investigations) | 0 | 1 | 0 — Non-Ocular

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/03/NCT04081103/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-10): https://cdn.clinicaltrials.gov/large-docs/03/NCT04081103/SAP_001.pdf